CLINICAL TRIAL: NCT03619265
Title: Evaluation of Activity Levels, Inflammatory Markers, and Overall Wellness. A Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Evaluation of Activity Levels, Inflammatory Markers, and Overall Wellness.
Acronym: 114-012
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NIS114012
Record Dates: First submitted 2018-07-10; First posted 2018-08-07 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Range of Motion

STUDY DESIGN:
Intervention Model Description: A double-blinded, randomized, placebo-controlled, parallel-arm clinical study design will be used.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prickly pear juice (Experimental): Prickly pear juice, 3 oz daily for 8 weeks.
  Interventions: Dietary Supplement: Prickly pear juice
- Pear-flavored juice (Placebo Comparator): Pear-flavored juice, 3 oz daily for 8 weeks.
  Interventions: Dietary Supplement: Pear-flavored juice

INTERVENTIONS:
Dietary Supplement: Prickly pear juice — 3 ounces daily for 8 weeks.
  Arms: Prickly pear juice
Dietary Supplement: Pear-flavored juice — 3 ounces daily for 8 weeks.
  Arms: Pear-flavored juice

SUMMARY:
The purpose for this protocol is to perform a double-blind, randomized, placebo-controlled, parallel-arm clinical study in healthy subjects to evaluate the efficacy of a nutraceutical product on physical and mental energy levels and overall wellness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of either gender;
* 35-75 years old;
* Chronic joint/muscle related pain for at least past 6 months;
* Body mass index (BMI) at or below 34.9 kg/m2.

Exclusion Criteria:

* Bariatric surgery;
* Diagnosed with diabetes Type I;
* Taking medication for diabetes Type II;
* Known serious chronic health condition;
* Serious active illness within past 12 months;
* Major surgery within the past 3 months;
* Major trauma within the past 3 months;
* Alcohol consumption of more than four standard units/day (for example more than four regular 12 oz beers (5% alcohol), four small 5-oz glasses of wine (12% alcohol), or four 1.5 oz shots of 80-proof spirits), or more than 28 units per week;
* Daily consumption of Nopalea or similar juice products during the past month;
* Currently taking anti-inflammatory nutritional supplements judged by the study coordinator to negate or camouflage the effects of the test product;
* Taking anti-inflammatory medications on a daily basis (81 mg aspirin is acceptable);
* Use of oral, inhaled or injected steroid medication within the last 6 months (for example: prednisone, dexamethasone). Nasal sprays for allergies are allowed;
* Any other significant disease or disorder that the investigator judges may put the subject at risk because of participation in the study, or may influence the result of the study;
* Any other condition or observation that the investigator judges may adversely affect the person's ability to complete the study;
* Women of child-bearing potential: Pregnant, breast-feeding, or trying to become pregnant;
* Known allergies to ingredients in the test and placebo products.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Pain level | Baseline, 2 weeks, and 8 weeks.
  Pain questionnaire: Scale 0-10, with 0 being pain-free and 10 being the most pain. Change from baseline will be evaluated.

SECONDARY OUTCOMES:
Range of motion | Baseline and 8 weeks.
  Digital inclinometry for measuring mobility of neck, back, hips, knees, and shoulders.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States